CLINICAL TRIAL: NCT03028090
Title: A Two-Arm Prospective, Multi-Centered Study to Assess Electrocardiogram Waveforms Produced Through the Utilization of the Sherlock 3CG™ Tip Confirmation System
Brief Title: Study to Assess Electrocardiogram Waveforms Produced Through the Utilization of the Sherlock 3CG™ Tip Confirmation System
Acronym: MODUS
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BAS-13-001
Record Dates: First submitted 2017-01-15; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Indication for Peripheral Intravenous Catheterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: SHERLOCK 3CG™ Tip Confirmation System with MODUS Software — The SHERLOCK 3CG™ Tip Confirmation System (TCS) is a fully-integrated magnetic tracking and ECG-based PICC tip confirmation technology. It was cleared by the FDA on March 19, 2012 and is indicated for use as an alternative to chest x-ray and fluoroscopy for PICC tip placement confirmation in adult patients. In order to further develop the SHERLOCK 3CG™ platform and simplify the PICC placement for the clinician, Bard Access Systems, Inc. is developing MODUS, a software package.

SUMMARY:
This study was to gather real-time ECG data through the use of the SHERLOCK 3CG™ Tip Confirmation System (TCS), an electrocardiogram (ECG)-based peripherally-inserted central catheter (PICC) tip confirmation technology. The study was to promote the development of a software package (MODUS) that can accurately define the maximum P-wave on an ECG waveform. All study participants received PICCs as their standard of care.

DETAILED DESCRIPTION:
The SHERLOCK 3CG™ Tip Confirmation System (TCS) is a fully integrated magnetic tracking and ECG-based PICC tip confirmation technology. It was cleared by the FDA on March 19, 2012 and is indicated for use as an alternative to chest x-ray and fluoroscopy for PICC tip placement confirmation in adult patients.

In order to further develop the SHERLOCK 3CG™ platform and simplify the PICC placement for the clinician, Bard Access Systems, Inc. developed a software package, MODUS, which can accurately define the maximum p-wave on an ECG waveform. This software provides visual and/or audio queues to notify the PICC placer of the location of the tip of the PICC relative to the cavoatrial junction of the patient.

Subjects who required bedside PICC placement as standard of care and met eligibility criteria were enrolled. The software package was not used in the guidance or placement of the PICC tip. PICCs were placed per standard of care procedure using anthropometric measurements with the SHERLOCK 3CG™ TCS System. Data from the placements was sent back to Bard for analysis.

ELIGIBILITY:
Inclusion Criteria:

A subject must have met the following criteria to be enrolled in the study:

1. Male or female, age ≥ 21 years
2. Subject required PICC placement as part of standard of care
3. Subject had signed an Informed Consent Form (ICF) or had an ICF signed by the subject's legally authorized representative

Exclusion Criteria:

* A subject was excluded if any of the following criteria were met:

  1. Subject had a contraindication to PICC placement as listed in the Instructions for Use (IFU)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was to be comprised of a sufficient number of subjects so that a minimum of 201 subjects completed the study, but no more than 250 subjects were to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percent agreement between maximum P-wave assessments of PICC nurse clinicians and the MODUS software during PICC insertion | The PICC insertion procedure is 60-90 mins in duration
  The measurement used will be percent agreement between clinician and MODUS software. Agreement of 95% between the nurse clinician and software assessments will be used to validate the study hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Gilbert, BSN, Study Director — CR Bard
Locations (2):
- United States (2):
  - Memorial Health System, Colorado Springs, Colorado
  - Bethesda North Hospital, Montgomery, Ohio